CLINICAL TRIAL: NCT02616185
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF ESCALATING DOSES OF A VACCINE-BASED IMMUNOTHERAPY REGIMEN (VBIR) FOR PROSTATE CANCER (PF-06753512)
Brief Title: A Phase 1 Study To Evaluate Escalating Doses Of A Vaccine-Based Immunotherapy Regimen For Prostate Cancer (PrCa VBIR)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to strategic evaluation of PF-06753512 (VBIR-1) within context of Pfizer's oncology portfolio, decision not based on any safety or regulatory concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B7791001; PRCA VBIR FIP STUDY (Other: Alias Study Number)
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation (Experimental): PF-06753512
  Interventions: Biological: PF-06755992; Biological: PF-06755990; Device: TDS-IM Electroporation Device; Biological: Tremelimumab; Biological: PF-06801591; Biological: PF-06753512

INTERVENTIONS:
Biological: PF-06755992 — PF-06755992 will be administered on Day 1 of Cycles 1 and 2.
  Other Names: AdC68
Biological: PF-06755990 — PF-06755990 will be administered using a device on Day 29, 57 and 85 of each cycle.
  Other Names: pDNA
Device: TDS-IM Electroporation Device — TDS-IM electroporation device and associated supplies will be used for PF-06755990 administration
Biological: Tremelimumab — PF-06753388 will be administered every 28 days.
  Other Names: PF-06753388
Biological: PF-06801591 — PF-06801591 will be administered every 28 days.
Biological: PF-06753512 — Combination of adenovirus (AdC68) + plasmid DNA (pDNA) + tremelimumab
  Other Names: VBIR-1 or PrCa VBIR

SUMMARY:
The study will evaluate the safety, pharmacokinetics and pharmacodynamics of increasing doses of a vaccine-based immunotherapy regimen for patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of prostate cancer
* Adequate bone marrow, kidney and liver function
* Hormone sensitive relapsing prostate cancer after definitive local therapy (biochemical relapse) OR
* Failed prior therapy with a novel hormone (e.g. enzalutamide, abiraterone) with documented progressive disease (post-novel hormone therapy CRPC)

Exclusion Criteria:

* ECOG performance status greater than or equal to 2
* Concurrent immunotherapy for prostate cancer
* History of or active autoimmune disorders (including but not limited to: myasthenia gravis, thyroiditis, pneumonitis, rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosus, scleroderma) and other conditions that disorganize or alter the immune system.
* History of inflammatory bowel disease.
* Current use of any implanted electronic stimulation device
* For biochemically relapsed patients, no concurrent use of ADT or orchiectomy and no known prior or current evidence of any metastatic involvement of distant organs
* For post-novel hormone patients, no concurrent treatment with a secondary hormone (e.g. enzalutamide, abiraterone), no metastasis to the liver or brain

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 91 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Banner-University Medical Center Tucson, Tucson, Arizona
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - GU Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Garden State Urology, Morristown, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Garden State Urology, Rockaway, New Jersey
  - Garden State Urology, Whippany, New Jersey
  - Northwell Health, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center 53rd Street, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, Sidney Kimmel Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Autio KA, Higano CS, Nordquist L, Appleman LJ, Zhang T, Zhu XH, Babiker H, Vogelzang NJ, Prasad SM, Schweizer MT, Madan RA, Billotte S, Cavazos N, Bogg O, Li R, Chan K, Cho H, Kaneda M, Wang IM, Zheng J, Tang SY, Hollingsworth R, Kern KA, Petrylak DP. First-in-human, phase 1 study of PF-06753512, a vaccine-based immunotherapy regimen (VBIR), in non-metastatic hormone-sensitive biochemical recurrence and metastatic castration-resistant prostate cancer (mCRPC). J Immunother Cancer. 2023 Mar;11(3):e005702. doi: 10.1136/jitc-2022-005702. PMID 36948505
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7791001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 123 participants were screened and 91 of them were assigned and treated in this study.
Groups:
- Cohort 1A: Adenovirus C68 (AdC68) 4x10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg: Participants with metastatic castrate resistant prostate cancer (mCRPC) in Cohort 1A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 4x10^11 VP Intramuscularly (IM) on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. Following the 2 cycles, participants in Cohort 1A entered the maintenance phase and received pDNA 5 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg: Participants with mCRPC in Cohort 2A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. Following the 2 cycles, participants in Cohort 2A entered the maintenance phase and received pDNA 5 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 80 mg: Participants with mCRPC in Cohort 3A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg was also administered subcutaneously (SC) after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 3A entered the maintenance phase and received pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg: Participants with mCRPC in Cohort 6A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg and PF-06801591 130 mg were also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 6A entered the maintenance phase and received PF-06801591 130 mg every month starting from Month 9, as well as pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg: Participants with mCRPC in Cohort 7A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg and PF-06801591 300 mg were also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 7A entered the maintenance phase and received PF-06801591 300 mg every month starting from Month 9, as well as pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg: Participants with mCRPC in Cohort 9A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 40 mg and PF-06801591 130 mg were also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 9A entered the maintenance phase and received PF-06801591 130 mg every month starting from Month 9, as well as pDNA 5 mg and tremelimumab 40 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg: Participants with biochemical relapse (BCR) of prostate cancer in Cohort 1B received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg was also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 1B entered the maintenance phase and received pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg: Participants with mCRPC in Cohort 3B received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg and PF-06801591 300 mg were also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 3B entered the maintenance phase and received PF-06801591 300 mg every month starting from Month 9, as well as pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg: Participants with BCR of prostate cancer in Cohort 5B received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg and PF-06801591 130 mg were also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 5B entered the maintenance phase and received PF-06801591 130 mg every month starting from Month 9, as well as pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
Period: Overall Study
Arm/Group | Cohort 1A: Adenovirus C68 (AdC68) 4x10^11 Viral Particles (VP) + Plasmid DNA (pDNA) 5 mg | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Tremelimumab (Treme) 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Started | 3 | 4 | 6 | 8 | 14 | 3 | 20 | 18 | 15
Completed | 2 | 3 | 3 | 3 | 5 | 2 | 12 | 5 | 9
Not Completed | 1 | 1 | 3 | 5 | 9 | 1 | 8 | 13 | 6
Not completed — Death | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 2 | 0
Not completed — Participant refused further follow-up | 1 | 1 | 2 | 3 | 4 | 0 | 3 | 4 | 3
Not completed — Not reported | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of one of the components of the regimen.
Groups:
- Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg: Participants with mCRPC in Cohort 1A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 4x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. Following the 2 cycles, participants in Cohort 1A entered the maintenance phase and received pDNA 5 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg: Participants with mCRPC in Cohort 3A received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg was also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 3A entered the maintenance phase and received pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg: Participants with BCR of prostate cancer in Cohort 1B received 2 repeated cycles (16 weeks each) of treatment, including AdC68 6x10^11 VP IM on Day 1 of Cycle 1 and 2, and pDNA 5 mg IM on Day 29, 57, and 85 of Cycle 1 and 2. On Day 1, 29, 57, and 85 of Cycle 1 and 2, tremelimumab 80 mg was also administered SC after the AdC68 or pDNA administration. Following the 2 cycles, participants in Cohort 1B entered the maintenance phase and received pDNA 5 mg and tremelimumab 80 mg every 2 months starting from Month 10, as long as there was clinical benefit.
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Total
Number analyzed (Participants) | 3 | 4 | 6 | 8 | 14 | 3 | 20 | 18 | 15 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 2 | 4 | 3 | 0 | 6 | 3 | 4 | 22
  >=65 years | 3 | 4 | 4 | 4 | 11 | 3 | 14 | 15 | 11 | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 4 | 6 | 8 | 14 | 3 | 20 | 18 | 15 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 4 | 6 | 8 | 14 | 3 | 18 | 17 | 15 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 6 | 7 | 12 | 2 | 19 | 13 | 13 | 79
  Black | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 4 | 2 | 11
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation where participant administered a product; the event did not need to have a causal relationship with the treatment. A SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to 6 months after End of Treatment (EOT; 52 months in maximum)
Population: Safety analysis set: all enrolled participants who received at least one dose of one of the components of the regimen. For this outcome measure, participants are grouped by disease type and treatment, as follows: Cohort All mCRPC Patients (all mCRPC participants), Cohort 1B (BCR with 1 immune checkpoint inhibitor [ICI]), Cohort 5B (BCR with 2 ICIs), and Cohort 7A and 3B Combined (mCRPC at recommended Phase 2 dose [RP2D] dose).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort All mCRPC Patients: This group included all mCRPC participants in the study (Cohort 1A, 2A, 3A, 6A, 7A, 9A, 3B).
- Cohort 7A and 3B Combined: This group included mCRPC participants in 7A and 3B, treated at RP2D dose.
Arm/Group | Cohort All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A and 3B Combined
Number analyzed (Participants) | 56 | 20 | 15 | 32
Participants
  Number of participants with all-causality AEs | 55 | 20 | 15 | 32
  Number of participants with treatment-related AEs | 51 | 19 | 15 | 31
  Number of participants with all-causality SAEs | 16 | 2 | 6 | 11
  Number of participants with treatment-related SAEs | 11 | 0 | 6 | 9

2. Primary Outcome: Number of Participants With AEs as Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03) (Grade >= 3)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. Grades of AEs were defined by NCI CTCAE v 4.03. Grade 1=asymptomatic/mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2=minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activity of daily living (ADL); Grade 3=severe or medically significant but not immediately life-threatening, hospitalization of prolongation of hospitalization indicated; disabling limiting self-care ADL; Grade 4=events with life-threatening consequences, urgent intervention indicated; Grade 5= death related to AE. Treatment-emergent adverse events occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 7A and 3B Combined: This group included mCRPC participants in 7A and 3B.
Arm/Group | Cohort All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A and 3B Combined
Number analyzed (Participants) | 56 | 20 | 15 | 32
Participants
  Grade 3 or Grade 4 (all-causality) | 33 | 10 | 11 | 21
  Grade 3 or Grade 4 (treatment-related) | 23 | 6 | 10 | 17
  Grade 5 (all-causality) | 4 | 0 | 1 | 3
  Grade 5 (treatment-related) | 1 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With AEs Leading to Discontinuation or Dose Reduction
Description: An AE was any untoward medical occurrence in a clinical investigation where participant administered a product; the event did not need to have a causal relationship with the treatment.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: Safety analysis set: all enrolled participants who received at least one dose of one of the components of the regimen. or this outcome measure, participants are grouped by disease type and treatment, as follows: Cohort All mCRPC Patients (all mCRPC participants), Cohort 1B (BCR with 1 immune checkpoint inhibitor [ICI]), Cohort 5B (BCR with 2 ICIs), and Cohort 7A and 3B Combined (mCRPC at recommended Phase 2 dose [RP2D] dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A and 3B Combined
Number analyzed (Participants) | 56 | 20 | 15 | 32
Participants
  Number of participants with permanent discontinuations | 16 | 1 | 10 | 11
  Number of participants with temporary discontinuations | 17 | 5 | 5 | 9
  Number of participants with dose reductions | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: The following AEs occurring in the first 28 days following the first AdC68 vaccination and not related to disease/progression were DLTs: (a) hematologic (Cohorts 1A to 3A and Cohorts 6A to 9A): Grade 3 neutropenia lasting >7 days, febrile neutropenia, Grade >=3 neutropenic infection, Grade >=3 thrombocytopenia, Grade >=3 anemia lasting >7 days, Grade >=3 lymphopenia lasting >14 days; (b) non-hematologic (all cohorts): Grade >=3 laboratory abnormalities either associated with symptoms or associated with worsening of an existing condition or that suggested a new disease process or that required additional active management, Grade >=3 toxicities, Grade 3 flu like symptoms lasting >3 days, fever of >40.0 degree Celsius lasting >3 days. Other clinically important or persistent toxicities at discretion of investigator and Pfizer.
Time Frame: The first 28 days following the first AdC68 vaccination (on Cycle 1 Day 1)
Population: Per protocol analysis set: all enrolled participants who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 and did not have major protocol deviations during the 28 days after the first vaccination. For this outcome measure, participants are grouped by disease type and treatment, as follows: Cohort All mCRPC Patients (all mCRPC participants), Cohort 1B (BCR with 1 ICI), Cohort 5B (BCR with 2 ICIs), and Cohort 7A and 3B Combined (mCRPC at RP2D dose).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort All mCRPC Patients: This group included all mCRPC participants in study (Cohort 1A, 2A, 3A, 6A, 7A, 9A, 3B).
Arm/Group | Cohort All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A and 3B Combined
Number analyzed (Participants) | 54 | 20 | 15 | 32
Participants | 1 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Hematology (Grade 3 or 4)
Description: Laboratory abnormalities were graded per NCI CTCAE version 4.03 (Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) and those with at least 1 participant are presented here. Hematology parameters included hemoglobin, platelets, white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: Safety analysis set: all enrolled participants who received at least one dose of one of the components of the regimen. For this outcome measure, participants are grouped by disease type and treatment, as follows: Cohort All mCRPC Patients (all mCRPC participants), Cohort 1B (BCR with 1 ICI), Cohort 5B (BCR with 2 ICIs), and Cohort 7A and 3B Combined (mCRPC at RP2D dose).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A and 3B Combined
Number analyzed (Participants) | 56 | 20 | 15 | 32
Participants
  Anemia | 2 | 0 | 0 | 2
  Hemoglobin increased | 0 | 0 | 0 | 0
  Lymphocyte count increased | 0 | 0 | 0 | 0
  Lymphopenia | 7 | 2 | 2 | 4
  Neutrophils (absolute) | 1 | 0 | 0 | 1
  Platelets | 0 | 0 | 0 | 0
  White blood cells | 1 | 0 | 0 | 1

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Chemistry (Grade 3 or 4)
Description: Laboratory abnormalities were graded per NCI CTCAE version 4.03 (Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) and those with at least 1 participant are presented here. Chemistry parameters included aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen (or urea), creatinine, uric acid, glucose, albumin, phosphorous or phosphate, lactate dehydrogenase, lipase, bicarbonate or carbon dioxide, total protein, TSH (if abnormal, reflex free T4 and free T3).
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- Cohort All mCRPC Patients: This group includes all mCRPC participants in study (Cohort 1A, 2A, 3A, 6A, 7A, 9A, 3B).
- Cohort 7A and 3B Combined: This group includes mCRPC participants in 7A and 3B.
Arm/Group | Cohort All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A and 3B Combined
Number analyzed (Participants) | 56 | 20 | 15 | 32
Participants
  Alanine aminotransferase | 1 | 0 | 1 | 0
  Alkaline phosphatase | 0 | 0 | 0 | 0
  Amylase | 2 | 0 | 0 | 0
  Aspartate aminotransferase | 1 | 0 | 1 | 0
  Bilirubin (total) | 0 | 1 | 0 | 0
  Creatinine | 1 | 0 | 0 | 0
  Hypercalcemia | 0 | 0 | 0 | 0
  Hyperglycemia | 4 | 0 | 0 | 2
  Hyperkalemia | 1 | 0 | 0 | 0
  Hypermagnesemia | 7 | 8 | 6 | 1
  Hypernatremia | 0 | 0 | 0 | 0
  Hypoalbuminemia | 0 | 0 | 0 | 0
  Hypocalcemia | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 0 | 0 | 0
  Hypokalemia | 3 | 0 | 0 | 2
  Hypomagnesemia | 0 | 0 | 0 | 0
  Hyponatremia | 0 | 1 | 2 | 0
  Hypophosphatemia | 2 | 5 | 4 | 1
  Lipase | 9 | 3 | 2 | 6

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Urinalysis (Grade 3 or 4)
Description: Laboratory abnormalities were graded per NCI CTCAE version 4.03 (Grade 3: severe AE; Grade 4: life-threatening consequences, urgent intervention indicated) and those with at least 1 participant are presented here. Urine parameters included urine protein and urine blood.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A and 3B Combined
Number analyzed (Participants) | 56 | 20 | 15 | 32
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in T Cell Response to Prostate Specific Antigen (PSA) in Part A
Description: T cell response to PSA was determined by assaying peripheral blood mononuclear cell (PBMC) samples for cellular immune responses against PSA antigens and was determined as the frequency of interferon-gamma (IFN-γ) spot forming cells (SFC)/million PBMCs. Change from baseline at Cycle 1 Day 71 and at Cycle 2 Day 99 are presented here.
Time Frame: At screening; Cycle 1: at Day 1, Day 15, Day 29, Day 43, Day 71; Cycle 2: at Day 1, Day 29, and Day 99; at the EOT visit, and 2, 4 and 6 months after EOT.
Population: All enrolled participants in Part A who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis. Number of Participants Analyzed = number of participants evaluable for this OM; Number Analyzed = number of participants evaluable for this OM at the time point specified.
Measure: Mean (Standard Deviation); unit: SFC/10^6 PBMCS
Arm/Group | Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 3 | 3 | 5 | 1 | 2 | 2
SFC/10^6 PBMCS
  Cycle 1 Day 1 Compared With Cycle 1 Day 71 | 2.83 (4.907) | 4.17 (7.217) | 1.70 (3.801) | NA (NA) — Titers were below the assay detection limit. | 24.25 (34.295) | NA (NA) — Titers were below the assay detection limit.
  Cycle 2 Day 1 Compared With Cycle 2 Day 99: number analyzed (Participants) | 2 | 3 | 2 | 0 | 0 | 0
  Cycle 2 Day 1 Compared With Cycle 2 Day 99 | NA (NA) — Titers were below the assay detection limit. | 5.50 (9.526) | NA (NA) — Titers were below the assay detection limit. |  |  |

9. Secondary Outcome: Change From Baseline in T Cell Response to Prostate Stem Cell Antigen (PSCA) in Part A
Description: T cell response to PSCA was determined by assaying PBMC samples for cellular immune responses against PSCA antigens and was determined as the frequency of IFN-γ SFC/million PBMCs. Change from baseline at Cycle 1 Day 71 and at Cycle 2 Day 99 are presented here.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: SFC/10^6 PBMCS
Arm/Group | Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 3 | 3 | 5 | 1 | 2 | 2
SFC/10^6 PBMCS
  Cycle 1 Day 1 Compared With Cycle 1 Day 71 | NA (NA) — Titers were below the assay detection limit. | NA (NA) — Titers were below the assay detection limit. | 1.70 (3.801) | NA (NA) — Titers were below the assay detection limit. | NA (NA) — Titers were below the assay detection limit. | NA (NA) — Titers were below the assay detection limit.
  Cycle 2 Day 1 Compared With Cycle 2 Day 99: number analyzed (Participants) | 2 | 3 | 2 | 0 | 0 | 0
  Cycle 2 Day 1 Compared With Cycle 2 Day 99 | NA (NA) — Titers were below the assay detection limit. | NA (NA) — Titers were below the assay detection limit. | NA (NA) — Titers were below the assay detection limit. |  |  |

10. Secondary Outcome: Change From Baseline in T Cell Response to Prostate Specific Membrane Antigen (PSMA) in Part A
Description: T cell response to PSMA was determined by assaying PBMC samples for cellular immune responses against PSMA antigens and was determined as the frequency of IFN-γ SFC/million PBMCs. Change from baseline at Cycle 1 Day 71 and at Cycle 2 Day 99 are presented here.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: SFC/10^6 PBMCS
Arm/Group | Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 3 | 3 | 5 | 1 | 2 | 2
SFC/10^6 PBMCS
  Cycle 1 Day 1 Compared With Cycle 1 Day 71 | 5.50 (9.526) | 28.00 (48.497) | 4.30 (12.736) | NA (NA) — Titers were below the assay detection limit. | NA (NA) — Titers were below the assay detection limit. | NA (NA) — Titers were below the assay detection limit.
  Cycle 2 Day 1 Compared With Cycle 2 Day 99: number analyzed (Participants) | 2 | 3 | 2 | 0 | 0 | 0
  Cycle 2 Day 1 Compared With Cycle 2 Day 99 | NA (NA) — Titers were below the assay detection limit. | 36.00 (62.354) | NA (NA) — Titers were below the assay detection limit. |  |  |

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tremelimumab in Part A
Description: Cmax was defined as the maximum observed plasma concentration. Blood samples (approximately 3 mL whole blood) to provide at least 1 mL of serum for measurement of tremelimumab PK analysis were collected.
Time Frame: Cycle 1: at Day 1 pre-dose, any time between 48 to 120 hr, approximately 168 hr, 336 hr, and 504 hr, at pre-dose on Day 29, Day 57, and Day 85; Cycle 2: at pre-dose on Day 1 and Day 29; at EOT visit, and 2, 4 and 6 months after EOT.
Population: All enrolled participants treated in Part A who had sufficient information to estimate at least 1 of the PK parameters of interest and who had no major protocol deviations influencing the PK assessment. Participants in Part 1 Cohort 3A, 6A, 7A, and 9A were treated with tremelimumab, thus included in this outcome measure. Summary statistics for Cohort 6A, 7A, and 9A are not presented since no participants had reportable parameter values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 6 | 0 | 0 | 0
ng/mL | 4360 (31) |  |  |

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Tremelimumab in Part A
Description: Tmax was defined as the time to reach maximum observed plasma concentration. Blood samples (approximately 3 mL whole blood) to provide at least 1 mL of serum for measurement of tremelimumab PK analysis were collected.
Time Frame: as for outcome 11
Population: All enrolled participants treated in Part A who had sufficient information to estimate at least 1 of the PK parameters of interest and who had no major protocol deviations influencing the PK assessment. Participants in Part 1 Cohort 3, 6, 7, and 9 were treated with tremelimumab, thus included in this outcome measure. Summary statistics for Cohort 6A, 7A, and 9A are not presented since no participants had reportable parameter values.
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 6 | 0 | 0 | 0
Hour | 307 [165 to 477] |  |  |

13. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Tremelimumab in Part A
Description: AUClast was defined as the area under the curve from time zero to last quantifiable concentration. Blood samples (approximately 3 mL whole blood) to provide at least 1 mL of serum for measurement of tremelimumab PK analysis were collected.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 6 | 0 | 0 | 0
ng*hr/mL | 2423000 (34) |  |  |

14. Secondary Outcome: Trough Concentrations (Ctrough) After Multiple Dosing of Tremelimumab
Description: Pre-dose tremelimumab concentration on Cycle 2 Day 1 is presented here as Ctrough. Blood samples (approximately 3 mL whole blood) to provide at least 1 mL of serum for measurement of tremelimumab PK analysis were collected. Summary statistics of Ctrough were not calculated if number of observations above lower lit of quantification (NALQ)=0 or <=3 participants had non-missing data.
Time Frame: Pre-dose on Cycle 2 Day 1
Population: PK parameter analysis population: all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest and who had no major protocol deviations influencing the PK assessment. Participants in Cohort 3A, 6A, 7A, 9A, 1B, 3B, and 5B were treated with tremelimumab, thus included in this outcome measure. Number of Participants Analyzed = Number of participants who had non-missing data and were evaluable for this OM.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 2 | 2 | 6 | 1 | 11 | 9 | 4
ng/mL | NA (NA) — Summary statistics were not computed for PK parameters when fewer than 3 participants had non-missing data. As per the statistical analysis plan of this study, data are considered not sufficient to calculate scientifically meaningful mean and standard deviation when sample size is less than 3. | NA (NA) — Summary statistics were not computed for PK parameters when fewer than 3 participants had non-missing data. As per the statistical analysis plan of this study, data are considered not sufficient to calculate scientifically meaningful mean and standard deviation when sample size is less than 3. | 5130 (1844.4) | NA (NA) — Summary statistics were not computed for PK parameters when fewer than 3 participants had non-missing data. As per the statistical analysis plan of this study, data are considered not sufficient to calculate scientifically meaningful mean and standard deviation when sample size is less than 3. | 4750 (2573.5) | 4849 (2726.7) | 5320 (1114.5)

15. Secondary Outcome: Cmax of PF-06801591 in Part A
Description: Cmax was defined as the maximum observed plasma concentration. Blood samples (approximately 5 mL) to provide serum for the analysis of PF-06801591 concentrations were collected.
Time Frame: as for outcome 11
Population: All enrolled participants treated in Part A who had sufficient information to estimate at least 1 of the PK parameters of interest and who had no major protocol deviations influencing the PK assessment. Participants in Part 1 Cohort 6A, 7A, and 9A were treated with PF-06801591, thus included in this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 8 | 14 | 3
ng/mL | 8507 (48) | 19960 (40) | 8899 (41)

16. Secondary Outcome: Tmax of PF-06801591 in Part A
Description: Tmax was defined as the time at which Cmax occurred. Blood samples (approximately 5 mL) to provide serum for the analysis of PF- 06801591 concentrations were collected.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 8 | 14 | 3
Hour | 164 [89.6 to 380] | 188 [67.3 to 378] | 166 [71.0 to 166]

17. Secondary Outcome: AUClast of PF-06801591 in Part A
Description: AUClast was defined as the area under the curve from time zero to last quantifiable concentration. Blood samples (approximately 5 mL) to provide serum for the analysis of PF-06801591 concentrations were collected. The geometric mean and geometric coefficient of variation of AUClast for Cohort 9A were not presented because fewer than 3 participants had reportable parameter values.
Time Frame: as for outcome 11
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg
Number analyzed (Participants) | 7 | 13 | 2
ng*hr/mL | 4095000 (43) | 10370000 (42) | NA (NA) — Fewer than 3 participants had reportable parameter values.

18. Secondary Outcome: Ctrough of PF-06801591
Description: Pre-dose PF-06801591 concentration on Cycle 2 Day 1 is presented here as Ctrough. Blood samples (approximately 3 mL whole blood) to provide at least 1 mL of serum for measurement of PF-06801591 PK analysis were collected.
Time Frame: Pre-dose on Cycle 2 Day 1
Population: PK parameter analysis population: all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest and who had no major protocol deviations influencing the PK assessment. Participants in Cohort 6A, 7A, 9A, 3B, and 5B were treated with PF-06801591, thus included in this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 2 | 6 | 1 | 10 | 4
ng/mL | NA (NA) — Summary statistics were not computed for PK parameters when fewer than 3 participants had non-missing data. As per the statistical analysis plan of this study, data are considered not sufficient to calculate scientifically meaningful mean and standard deviation when sample size is less than 3. | 6873 (9097.8) | NA (NA) — Summary statistics were not computed for PK parameters when fewer than 3 participants had non-missing data. As per the statistical analysis plan of this study, data are considered not sufficient to calculate scientifically meaningful mean and standard deviation when sample size is less than 3. | 20880 (12114) | 3472 (5085.7)

19. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Against Tremelimumab
Description: Blood samples (approximately 5 mL) to provide at least 1 mL of serum to detect ADA were collected from participants enrolled in to Cohorts 3A to 9A and Cohorts 1B to 5B. Participants were considered ADA-positive if sample titer (log10) >=1.48; participants were considered ADA-negative if sample titer (log10) <1.48.
Time Frame: Cycle 1: at Day 1, Day 29, and Day 85; Cycle 2: at Day 29; at the EOT visit, and 2, 4 and 6 months after EOT. Samples collected on dosing days were obtained within 6 hours prior to tremelimumab dosing.
Population: All enrolled participants who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis. For this outcome measure, participants are grouped by disease type and tremelimumab dose, as follows: All mCRPC Patients, All BCR Patients, Cohort 9A (tremelimumab 40 mg), and Cohort 3A, 6A, 7A, 1B, 3B, and 5B Combined (tremelimumab 80 mg).
Measure: Count of Participants; unit: Participants
Groups:
- All mCRPC Patients: This group included all mCRPC participants in study who received tremelimumab (Cohort 3A, 6A, 7A, 9A, 3B).
- All BCR Patients: This group included all BCR participants in study who received tremelimumab (Cohort 1B and 5B).
- Cohort 3A, 6A, 7A, 1B, 3B and 5B Combined: This group included participants in 3A, 6A, 7A, 1B, 3B and 5B who received tremelimumab 80 mg.
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 3A, 6A, 7A, 1B, 3B and 5B Combined
Number analyzed (Participants) | 49 | 35 | 3 | 81
Participants | 6 | 11 | 1 | 16

20. Secondary Outcome: Titer of Treatment-Induced ADA Against Tremelimumab
Description: Treatment-induced ADA was defined as baseline titer missing or negative and participant had >=1 post-treatment positive titer. Blood samples (approximately 5 mL) to provide at least 1 mL of serum to detect ADA were collected from participants enrolled in to Cohorts 3A to 9A and Cohorts 1B to 5B.
Time Frame: as for outcome 19
Population: All enrolled participants who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis. For this outcome measure, participants are grouped by disease type and tremelimumab dose as follows: All mCRPC Patients, All BCR Patients, Cohort 9A (tremelimumab 40 mg), and Cohort 3A, 6A, 7A, 1B, 3B, and 5B Combined (tremelimumab 80 mg).
Measure: Median (Inter-Quartile Range); unit: 1/dilution
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 3A, 6A, 7A, 1B, 3B and 5B Combined
Number analyzed (Participants) | 6 | 11 | 1 | 16
1/dilution | 2.81 [2.68 to 2.91] | 2.34 [2.15 to 2.79] | 2.68 [2.68 to 2.68] | 2.70 [2.20 to 2.87]

21. Secondary Outcome: Number of Participants With Neutralizing Antibody (NAb) Against Tremelimumab
Description: Only those samples tested positive for ADA were to be further tested for Nab. Blood samples (approximately 5 mL) to provide at least 1 mL of serum to detect NAb were collected from participants enrolled in to Cohorts 3A to 9A and Cohorts 1B to 5B. Nab against tremelimumab was not examined due to business reason.
Time Frame: as for outcome 19
Population: as for outcome 20
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 3A, 6A, 7A, 1B, 3B and 5B Combined
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Titer of Treatment-Induced NAb Against Tremelimumab
Description: as for outcome 21
Time Frame: as for outcome 19
Population: as for outcome 20
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 3A, 6A, 7A, 1B, 3B and 5B Combined
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With ADA Against PF-06801591
Description: Participants were considered ADA-positive if sample titer (log10) >=99; Participants were considered ADA-negative if sample titer (log10) <99. Blood samples (approximately 5 mL) to provide at least 1 mL of serum for detection of ADA against PF-06801591 were collected from participants enrolled in Cohorts 6A to 9A and Cohorts 3B and 5B.
Time Frame: Cycle 1: at Day 1, Day 29, and Day 85; Cycle 2: at Day 29; at the EOT visit, and 2, 4 and 6 months after EOT. Samples collected on dosing days were obtained within 6 hours prior to PF-06801591 dosing.
Population: All enrolled participants who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis. For this outcome measure, participants are grouped by disease type and PF-06801591 dose as follows: All mCRPC Patients, All BCR Patients, Cohort 7A and 3B Combined (PF-06801591 300 mg), and Cohort 6A, 9A, and 5B Combined (PF-06801591 130 mg).
Measure: Count of Participants; unit: Participants
Groups:
- All mCRPC Patients: This group included all mCRPC participants in study who received PF-06801591 (Cohort 6A, 7A, 9A, and 3B).
- All BCR Patients: This group included all BCR participants in study who received PF-06801591 (Cohort 5B).
- Cohort 7A and 3B Combined: This group included mCRPC participants in 7A and 3B, who received PF-06801591 300 mg.
- Cohort 6A, 9A, and 5B Combined: This group included participants in 6A, 9A, and 5B, who received PF-06801591 130 mg.
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 7A and 3B Combined | Cohort 6A, 9A, and 5B Combined
Number analyzed (Participants) | 43 | 15 | 32 | 26
Participants | 5 | 8 | 3 | 10

24. Secondary Outcome: Titer of Treatment-Induced ADA Against PF-06801591
Description: Treatment-induced ADA was defined as baseline titer missing or negative and participant had >=1 post-treatment positive titer. Blood samples (approximately 5 mL) to provide at least 1 mL of serum for detection of ADA against PF-06801591 were collected from participants enrolled in Cohorts 6A to 9A and Cohorts 3B and 5B.
Time Frame: as for outcome 23
Population: All enrolled participants who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis. For this outcome measure, participants are grouped by disease type and PF-06801591 dose, as follows: All mCRPC Patients, All BCR Patients, Cohort 7A and 3B Combined (PF-06801591 300 mg), and Cohort 6A, 9A, and 5B Combined (PF-06801591 130 mg).
Measure: Median (Inter-Quartile Range); unit: 1/dilution
Groups:
- All mCRPC Patients: This group included all mCRPC participants in study who received PF-06801591(Cohort 6A, 7A, 9A, and 3B).
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 7A and 3B Combined | Cohort 6A, 9A, and 5B Combined
Number analyzed (Participants) | 5 | 6 | 3 | 8
1/dilution | 880 [790 to 16800] | 2010 [797 to 5070] | 790 [99 to 16800] | 2010 [838.5 to 6295]

25. Secondary Outcome: Number of Participants With NAb Against PF-06801591
Description: Only those samples tested positive for ADA were to be further tested for Nab. Blood samples (approximately 5 mL) to provide at least 1 mL of serum for detection of NAb against PF-06801591 were collected from participants enrolled in Cohorts 6A to 9A and Cohorts 3B and 5B. Nab against PF-06801591 was not examined due to business reason.
Time Frame: as for outcome 23
Population: as for outcome 24
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 7A and 3B Combined | Cohort 6A, 9A, and 5B Combined
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Secondary Outcome: Titer of Treatment-Induced NAb Against PF-06801591
Description: as for outcome 25
Time Frame: as for outcome 23
Population: as for outcome 24
Arm/Group | All mCRPC Patients | All BCR Patients | Cohort 7A and 3B Combined | Cohort 6A, 9A, and 5B Combined
Number analyzed (Participants) | 0 | 0 | 0 | 0

27. Secondary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Cohort 7A and 3B Combined and All mCRPC Patients
Description: ORR was defined as the percentage of participants with best overall response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST v1.1. Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm) and no new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease and no new lesions.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: All enrolled participants in Cohort 1A, 2A, 3A, 6A, 7A, 9A, and 3B who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All mCRPC Patients: This group included all mCRPC participants in study (Cohort 1A, 2A, 3A, 6A, 7A, 9A, and 3B).
Arm/Group | Cohort 7A and 3B Combined | All mCRPC Patients
Number analyzed (Participants) | 32 | 54
Percentage of participants | 9.4 [2.0 to 25.0] | 5.6 [1.2 to 15.4]

28. Secondary Outcome: Duration of Response (DOR) by RECIST v1.1 in Cohort 7A and 3B Combined and All mCRPC Patients
Description: DOR was defined as the time from first documentation of confirmed CR or PR to date of first documentation of progressive disease (PD) or death due to any cause according to RECIST v1.1. Per RECIST v1.1: CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm) and no new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all measurable target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease and no new lesions. PD was defined as >=20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. Unequivocal progression of pre existing lesions for non-target disease.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: as for outcome 27
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 7A and 3B Combined | All mCRPC Patients
Number analyzed (Participants) | 3 | 3
Days | 169 [119 to 224] | 169 [119 to 224]

29. Secondary Outcome: Immune-Related Confirmed ORR by Immune Related Response Evaluation Criteria in Solid Tumors Version 1.1 (irRECIST v1.1) in Cohort 7A and 3B Combined and All mCRPC Patients
Description: Immune-related confirmed ORR was defined as the percentage of participants with objective response based assessment of confirmed immune related complete response (irCR) or confirmed immune related partial response (irPR) according to irRECIST v1.1. Per irRECIST v1.1: irCR was defined as complete disappearance of all lesions and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 mm. irPR was defined as sum of the diameters (longest for non nodal lesions, shortest for nodal lesions) of target and new measurable lesions must decrease >=30%.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 7A and 3B Combined | All mCRPC Patients
Number analyzed (Participants) | 32 | 54
Percentage of participants | 9.4 [2.0 to 25.0] | 5.6 [1.2 to 15.4]

30. Secondary Outcome: Immune-Related Confirmed DOR by irRECIST v1.1 in Cohort 7A and 3B Combined and All mCRPC Patients
Description: Immune-related confirmed DOR was defined as the time from first documentation of confirmed irCR or confirmed irPR to date of first documentation of immune related progressive disease (irPD) or death due to any cause according to irRECIST. Per irRECIST v1.1: irCR was defined as complete disappearance of all lesions and no new lesions. All measurable lymph nodes also must have a reduction in short axis to <10 mm. irPR was defined as sum of the diameters (longest for non nodal lesions, shortest for nodal lesions) of target and new measurable lesions must decrease >=30%. irPD was defined as sum of the diameters of target and new measurable lesions must increase >=20%, confirmed by a repeat, consecutive observation at least 4 weeks from the date first documented.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: as for outcome 27
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 7A and 3B Combined | All mCRPC Patients
Number analyzed (Participants) | 3 | 3
Days | 169 [119 to 224] | 169 [119 to 224]

31. Secondary Outcome: Number of Patients With Bone Progression Per Prostrate Cancer Working Group 3 (PCWG3) Criteria in Cohort 7A and 3B Combined
Description: Number of participants with bone progression per Prostate Cancer Clinical Trials Working Group 3 (PCWG3). Per PCWG3, progressing disease on bone scan was considered when at least two new lesions relative to the first post treatment scan was confirmed on a subsequent scan (6 or more weeks later).
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: All enrolled participants in Cohort 7A and 3B who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 7A and 3B Combined
Number analyzed (Participants) | 32
Participants | 2

32. Secondary Outcome: Radiographic Progression Free Survival (rPFS) Per RECIST v1.1 in Cohort 7A and 3B Combined , All mCRPC Patients, Cohort 1B, and Cohort 5B
Description: Radiographic Progression Free Survival (rPFS) per RECIST v1.1. rPFS was defined as the time from first dose of study treatment to date of first documentation of radiographic PD or death due to any cause, whichever occurs first. Per RECIST v1.1, PD was defined as >=20% increase in the sum of diameters of target measurable lesions above the smallest sum observed, with a minimum absolute increase of 5 mm. Unequivocal progression of pre existing lesions for non-target disease. The Kaplan Meier estimate of median rPFS was presented here.
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Population: All enrolled participants who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 7A and 3B Combined | All mCRPC Patients | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 32 | 54 | 20 | 15
Months | 5.6 [2.0 to NA] — Not estimable based on Based on the Brookmeyer and Crowley method. | 5.6 [3.5 to NA] — Not estimable based on Based on the Brookmeyer and Crowley method. | NA [10.2 to NA] — Not estimable based on Based on the Brookmeyer and Crowley method. | NA [NA to NA] — Not estimable based on Based on the Brookmeyer and Crowley method.

33. Secondary Outcome: Number of Participants Achieving Central PSA Response >= 50% Decline From Baseline (PSA-50) in Part B
Description: PSA-50 response rate was defined as the proportion of patients whose on-study PSA declined from baseline by at least 50% at two consecutive measurements at least 3 weeks apart, prior to other systematic anti-cancer therapy.
Time Frame: At screening; Cycle 1 and 2: at Day 1, Day 29, Day 57, and Day 85; at the EOT visit, and 1, 2, 4 and 6 months after EOT.
Population: All enrolled participants in Part B who received at least one dose of all assigned regimen components administered on Cycle 1 Day 1 of treatment and must have at least 1 valid and determinate assay result related to the proposed analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 18 | 15
Participants | 5 | 1 | 3

34. Secondary Outcome: Duration of PSA-50 Response in Part B
Description: Duration of PSA-50 response was defined as the period from the first measurement when PSA-50 response was achieved to the measurement when PSA-50 response no longer held.
Time Frame: Days 1, 29, 57 of Cycle 1 and Cycle 2.
Population: as for outcome 33
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 5 | 1 | 3
Months | 6.9 [1.4 to 12.9] | 5.6 [5.6 to 5.6] | 4.1 [2.7 to 6.7]

35. Secondary Outcome: Baseline for PSA in Part B
Description: PSA Baseline is defined as the most recent non-missing value prior to dosing.
Time Frame: At screening and Cycle 1 Day 1.
Population: All enrolled participants in Part B who received at least one dose of one of the components of the regimen.
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 18 | 15
ng/ml
  Central PSA | 3.05 [1.8 to 20.1] | 33.45 [0.8 to 2136.0] | 2.10 [0.5 to 11.5]
  Local PSA | 3.050 [1.80 to 20.57] | 37.150 [0.70 to 1500.00] | 2.080 [0.50 to 12.43]

36. Secondary Outcome: Baseline for PSA Doubling Time (PSADT) in Part B
Description: PSADT was defined as the natural log of 2 divided by the slope of the linear regression line of the natural log of PSA against time in month. Baseline has been calculated from the PSA values at screening and C1D1.
Time Frame: At screening and Cycle 1 Day 1.
Population: as for outcome 33
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 13 | 12
Months | 1.768 [-10.04 to 7.73] | 1.169 [-78.50 to 11.82] | 1.615 [-10.28 to 20.72]

37. Secondary Outcome: Baseline for PSA Slope in Part B
Description: PSA slope was defined as the slope of the linear regression line of natural log of PSA against time in month. Baseline has been calculated from the PSA values at screening and C1D1.
Time Frame: At screening and Cycle 1 Day 1.
Population: as for outcome 33
Measure: Median (Full Range); unit: Ratio
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 13 | 12
Ratio | 0.178 [-0.20 to 0.75] | 0.205 [-0.31 to 0.73] | 0.138 [-0.28 to 0.47]

38. Secondary Outcome: Baseline for PSA Velocity in Part B
Description: PSA velocity was defined as the slope of the linear regression line of PSA against time in month. Baseline has been calculated from the PSA values at screening and C1D1.
Time Frame: At screening and Cycle 1 Day 1.
Population: as for outcome 33
Measure: Median (Full Range); unit: ng/ml/month
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 13 | 12
ng/ml/month | 0.558 [-0.87 to 6.67] | 3.629 [-63.41 to 46.04] | 0.109 [-1.24 to 0.91]

39. Secondary Outcome: Change in PSADT at Post-Treatment Visit From Baseline in Part B
Description: PSADT was defined as the natural log of 2 divided by the slope of the linear regression line of the natural log of PSA against time in month. PSADT at the post-treatment visit was calculated from C1D1 and all post-treatment PSA values.
Time Frame: At screening; Cycle 1 and 2: at Day 1, Day 29, Day 57, and Day 85; at the EOT visit, and 1, 2, 4 and 6 months after EOT.
Population: as for outcome 33
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 13 | 12
Months | 4.800 [-31.92 to 44.66] | 4.243 [-0.23 to 80.68] | 8.078 [-58.53 to 23.27]

40. Secondary Outcome: Change in PSA Slope at Post-Treatment Visit From Baseline in Part B
Description: PSA slope was defined as the slope of the linear regression line of natural log of PSA against time in month. PSA slope at the post-treatment visit was calculated from C1D1 and all post-treatment PSA values.
Time Frame: At screening; Cycle 1 and 2: at Day 1, Day 29, Day 57, and Day 85; at the EOT visit, and 1, 2, 4 and 6 months after EOT.
Population: as for outcome 33
Measure: Median (Full Range); unit: Ratio
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 13 | 12
Ratio | -0.084 [-0.68 to 0.97] | -0.067 [-0.38 to 0.70] | 0.076 [-0.61 to 0.34]

41. Secondary Outcome: Change in PSA Velocity at Post-Treatment Visit From Baseline in Part B
Description: PSA velocity was defined as the slope of the linear regression line of PSA against time in month. PSA velocity at the post-treatment visit was calculated from C1D1 and all post-treatment PSA values.
Time Frame: At screening; Cycle 1 and 2: at Day 1, Day 29, Day 57, and Day 85; at the EOT visit, and 1, 2, 4 and 6 months after EOT.
Population: as for outcome 33
Measure: Median (Full Range); unit: ng/ml/month
Arm/Group | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
Number analyzed (Participants) | 20 | 13 | 12
ng/ml/month | -0.008 [-4.50 to 5.46] | 8.641 [-9.56 to 473.67] | 0.185 [-0.58 to 2.30]

ADVERSE EVENTS:
Time Frame: Baseline up to 6 months after EOT (52 months in maximum)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AE reporting, including suspected unexpected serious adverse reactions, was carried out in accordance with applicable local regulations.
Arm/Group | Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/6 | 1/8 | 2/14 | 0/3 | 0/20 | 2/18 | 1/15
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 2/6 | 2/8 | 4/14 | 1/3 | 2/20 | 7/18 | 6/15
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 5/6 | 8/8 | 14/14 | 3/3 | 20/20 | 18/18 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg (N=3) | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg (N=4) | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg (N=6) | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg (N=8) | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg (N=14) | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg (N=3) | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg (N=20) | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg (N=18) | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg (N=15)
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immune-mediated myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 (0) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1A: AdC68 4x10^11 VP + pDNA 5 mg (N=3) | Cohort 2A: AdC68 6x10^11 VP + pDNA 5 mg (N=4) | Cohort 3A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg (N=6) | Cohort 6A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg (N=8) | Cohort 7A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg (N=14) | Cohort 9A: AdC68 6x10^11 VP + pDNA 5 mg + Treme 40 mg + PF-06801591 130 mg (N=3) | Cohort 1B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg (N=20) | Cohort 3B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 300 mg (N=18) | Cohort 5B: AdC68 6x10^11 VP + pDNA 5 mg + Treme 80 mg + PF-06801591 130 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 5 | 4 | 0 | 0 | 14 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 6 | 0 | 2 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 5 | 0 | 5 | 8 | 8
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 4 | 5 | 2 | 3 | 5 | 5
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 2 | 0 | 3 | 4 | 1
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Chills (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 5 | 2
Fatigue (General disorders) | 1 | 2 | 1 | 4 | 5 | 3 | 12 | 7 | 8
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Influenza like illness (General disorders) | 2 | 1 | 1 | 1 | 6 | 0 | 12 | 1 | 5
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discomfort (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2
Injection site reaction (General disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 2 | 1 | 0 | 4 | 3 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 (3) | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 4 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 3 | 5
Amylase increased (Investigations) | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 6 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 3 | 1
Blood pressure increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 1 | 3 | 0 | 5 | 6 | 5
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 4 | 4 | 1 | 2 | 6 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 3 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 3 | 0 | 1 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 4 | 6 | 2 | 8 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 3 | 1 | 5 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 5 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1 | 2 | 5 | 3 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 4 | 2
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 6 | 5 | 6
Hypersomnia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 3 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 4 | 1 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 4 | 2
Bladder neck obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 3 | 6 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 3 | 4
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 3 | 4
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 (1) | 3
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 6 | 2 | 3
Malaise (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 5 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 5 | 7
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 6 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 4
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 7 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 8 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 5 | 2
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 4 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 4 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thyroxine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0/7 | 0 | 0 | 0 | 0 | 1
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0/7 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated on 20 August 2020 by the sponsor. The decision to terminate this study was based on the results of a strategic evaluation of VBIR-1 within the current Pfizer oncology portfolio. This decision was not based on any safety or regulatory concerns with the treatment of participants with VBIR-1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT02616185/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT02616185/SAP_001.pdf